CLINICAL TRIAL: NCT00470470
Title: A Phase II Study of Imatinib Mesylate (STI571;NSC#716051:IND 61135) in Patients With Inoperable AJCC Stage III or IV Melanoma Harboring Somatic Alterations of C-KIT
Brief Title: Imatinib Mesylate in Treating Patients With Stage III or Stage IV Melanoma That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00216; NCI-2009-00216 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000543404; MSKCC-07014; 07-014 (Other: Memorial Sloan-Kettering Cancer Center); 7754 (Other: CTEP); P30CA008748 (NIH); N01CM62206 (NIH); N01CM62204 (NIH)
Record Dates: First submitted 2007-05-03; First posted 2007-05-07 (Estimated); Results first posted 2014-12-23 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-01

CONDITIONS: Acral Lentiginous Malignant Melanoma; Recurrent Melanoma; Stage IIIA Melanoma; Stage IIIB Melanoma; Stage IIIC Melanoma; Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — Imatinib Mesylate

ARMS (1):
- Treatment (enzyme inhibitor therapy) (Experimental): Patients receive oral imatinib mesylate twice daily for up to 12 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: imatinib mesylate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: imatinib mesylate — Given orally
  Other Names: CGP 57148; Gleevec; Glivec
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well imatinib mesylate works in treating patients with stage III or stage IV melanoma that cannot be removed by surgery. Imatinib mesylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the overall objective response rate (complete response and partial response) in patients with inoperable stage III or IV melanoma harboring somatic alterations in c-KIT treated with imatinib mesylate.

SECONDARY OBJECTIVES:

I. Determine the time to progression in patients treated with this drug. II. Determine if c-KIT mutational status by DNA sequencing, DNA copy number status by fluorescent in situ hybridization (FISH) or comparative genomic hybridization, and/or protein expression by immunohistochemistry (IHC) can best predict clinical benefit from imatinib mesylate.

TERTIARY OBJECTIVES:

I. To evaluate tumors resistant to small molecule inhibitors of Kit for the development of secondary Kit mutations or for changes in Kit copy number.

II. To evaluate for changes in Ki-67, phospho-Akt, phospho-MEK, phospho-S6, phospho STAT3, cleaved caspase 3, IGF-1R, and Kit expression in paired tumor samples obtained from patients treated with a small molecule inhibitor of Kit.

III. To analyze baseline and post-resistance blood samples for soluble cKIT levels, soluble VEGFR1, soluble VEGFR2, VEGF, PlGF, FGF, and melanoma inhibitory activity (MIA) levels, and circulating tumor cells.

IV. To analyze concomitant samples of blood and tumor for imatinib levels in patients treated with imatinib.

OUTLINE: This is a multi-center study. Patients are stratified according to true amplification of c-KIT by FISH vs mutations by DNA sequencing.

Patients receive oral imatinib mesylate twice daily for up to 12 weeks in the absence of disease progression or unacceptable toxicity.

Tumor tissue samples or unstained tissue slides/paraffin blocks may be collected. c-KIT is evaluated by IHC and comparative genomic hybridization.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed inoperable stage III or IV melanoma that began on acral skin or mucosa

  * Patients with cutaneous melanoma that began on sun exposed sites of the skin and whose pathology demonstrates signs of sun damage (solar elastosis) involving the skin surrounding their primary melanoma are eligible
* Must have sufficient tumor tissue available for FISH and DNA sequencing

  * Patients must have either a true amplification of 4q12 or a detectable mutation of c-KIT
  * If no banked tumor tissue is available, or if the available banked tumor tissue is insufficient for the necessary testing, then a repeat biopsy procedure will be required to collect the necessary tumor sample
* Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* No known untreated brain or epidural metastases

  * Brain metastases that have been treated and deemed stable are allowed
* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* Life expectancy greater than 3 months
* WBC ≥ 3,000/mm³
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)

  * Patients with unexplained hyperbilirubinemia that is clinically consistent with an inherited disorder of bilirubin metabolism (e.g., Gilbert's syndrome) may be eligible
* AST and ALT ≤ 2.5 times ULN (5 times ULN if hepatic metastases are present)
* Creatinine ≤ 1.5 times ULN
* PT and PTT ≤ 1.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception before and during study participation
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to imatinib mesylate
* No concurrent uncontrolled illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable anginapectoris
  * Cardiac arrhythmia resulting in hemodynamic instability
  * Intestinal malabsorption disorders
  * Psychiatric illness or social situations that would limit study compliance
* Recovered to grade 1 from all prior therapies with the exception of alopecia
* At least 2 weeks since prior radiotherapy (≤ 3,000 cGy to fields including substantial marrow)
* At least 2 weeks since prior isolated limb infusion or perfusion (must have evidence of progression despite this therapy)
* At least 2 weeks since prior chemotherapy
* No more than 2 prior chemotherapy regimen for metastatic melanoma
* Prior therapies with vaccines, targeted agents not believed to affect the kit proteins, cytokines, interferon-α, or intratumoral injections will NOT be considered prior therapy unless administered with a chemotherapy drug
* No prior therapy with an inhibitor of the kit protein
* No other concurrent investigational agents
* No other concurrent anticancer agents or therapies
* No concurrent antiretroviral therapy for HIV-positive patients
* No concurrent inhibitors of CYP3A4, including any of the following:

  * Fluconazole, itraconazole, ketoconazole, macrolide antibiotics (azithromycin, clarithromycin, erythromycin, troleandomycin),midazolam, nifedipine, verapamil, diltiazem, terfenadine, cyclosporine and cisapride
  * Herbal extracts and tinctures with CYP3A4 inhibitory activity, including the following:

    * Hydrastis canadensis (goldenseal), Hypericum perforatum (St. John's wort),Uncaria tomentosa (cat's claw), Echinacea angustifolia roots, Trifolium pratense(wild cherry), Matricaria, chamomilla (chamomile), Glycyrrhiza glabra (licorice), dillapiol, hypericin, and naringenin
* No concurrent inducers of CYP3A4, including any of the following:

  * Carbamazepine, phenobarbital, phenytoin, and rifampin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-04; Primary Completion 2013-12 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Carvajal, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - University of California at Los Angeles (UCLA ), Los Angeles, California
  - Mount Sinai Medical Center CCOP, Miami Beach, Florida
  - Good Samaritan Medical Center, West Palm Beach, Florida
  - Palm Beach Cancer Institute-Main Office, West Palm Beach, Florida
  - New York University Langone Medical Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York

REFERENCES:
- [Derived] Carvajal RD, Antonescu CR, Wolchok JD, Chapman PB, Roman RA, Teitcher J, Panageas KS, Busam KJ, Chmielowski B, Lutzky J, Pavlick AC, Fusco A, Cane L, Takebe N, Vemula S, Bouvier N, Bastian BC, Schwartz GK. KIT as a therapeutic target in metastatic melanoma. JAMA. 2011 Jun 8;305(22):2327-34. doi: 10.1001/jama.2011.746. PMID 21642685

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual: 04/05/2007
  Protocol Closed to Accrual: 11/23/2010
  Recruitment Location is the medical clinic
Groups:
- Treatment (Enzyme Inhibitor Therapy): Patients receive oral imatinib mesylate 400 mg twice daily for up to 12 weeks in the absence of disease progression or unacceptable toxicity.
  imatinib mesylate: Given orally
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Started | 30
Completed | 25
Not Completed | 5
Not completed — Adverse Event | 2
Not completed — Death | 2
Not completed — Not treated | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 30
Age, Continuous [Median (Standard Deviation); unit: years] | 68.5 (27.57716447)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Response will be evaluated in this study using the new international criteria proposed by the RECIST Committee. A Simon two-stage minimax design will be employed.
Time Frame: Every 6 weeks for the first 3 courses and then every 12 weeks thereafter
Measure: Number; unit: participants
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 25
participants
  Complete Response | 1
  Partial Response | 3
  Stable Disease | 14
  Progression of Disease | 7

2. Secondary Outcome: Time to Progression
Description: Progression will be evaluated in this study using the new international criteria proposed by the RECIST Committee. Time to progression will be estimated using the Kaplan-Meier method.
Time Frame: Time from the treatment start to the date of disease progression
Measure: Mean (Inter-Quartile Range); unit: weeks
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 25
weeks | 12 [6 to 18]

ADVERSE EVENTS:
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Serious Adverse Events (participants affected / at risk) | 18/30
Other Adverse Events (participants affected / at risk) | 23/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Enzyme Inhibitor Therapy) (N=30)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Serum amylase increased (Investigations) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Creatinine increased (Investigations) | 3 (3)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1)
Death (Disease progression) (General disorders) | 6 (6)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Edema (Head and Neck) (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Gynecomastia (Reproductive system and breast disorders) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 4 (4)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Hemorrhage-urinary tract (Renal and urinary disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Infection-Urinary tract (Infections and infestations) | 1 (1)
Lipase increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 3 (3)
Nausea (Gastrointestinal disorders) | 5 (5)
Obstruction-Ureter (Renal and urinary disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Platelet count decreased (Investigations) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 1 (1)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Enzyme Inhibitor Therapy) (N=30)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 13 (93)
Creatinine increased (Investigations) | 2 (15)
Edema-limbs (General disorders) | 2 (2)
Fatigue (General disorders) | 8 (9)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (5)
Hyponatremia (Metabolism and nutrition disorders) | 3 (8)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (6)
Lymphocyte count decreased (Investigations) | 7 (27)
Nausea (Gastrointestinal disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (8)
White blood cell decreased (Investigations) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less